CLINICAL TRIAL: NCT04336761
Title: Prevalence of Covid-19 in Children Admitted to Paediatric Emergency Departments During the Pandemic Period in France
Acronym: INCOVPED
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_21; 2020-A00811-38 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Coronavirus; COVID; Infection Viral
Keywords: pediatric emergencies; pandemia
MeSH Terms: conditions — Coronavirus Infections; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasopharyngeal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Child suspected of infection with COVID-19.: Child included with positive included
  Interventions: Diagnostic Test: nasopharyngeal swab

INTERVENTIONS:
Diagnostic Test: nasopharyngeal swab — Data collection and nasopharyngeal swab

SUMMARY:
Arriving in December 2019, Coronavirus COVID-19 infection is causing a global pandemic with high morbidity and mortality among adults and especially seniors. The child appears little or no affected by this infection. It is estimated that the child could be asymptomatic or pauci-symptomatic carrier and thus be vector of the disease. For this reason, measures have been taken to close schools and contain populations in a large number of countries, including France. However, there are no data on the prevalence of COVID-19 in children.

ELIGIBILITY:
Inclusion Criteria:

* 1st Line Consultation in Pediatric Emergencies
* All reasons for consultation during working hours
* Informed and written consent of a parent holder (only 1 authorized companion) and a child of understanding age

Exclusion Criteria:

* Refusal of participation by parents/child of decision age
* No membership of a social security scheme (beneficiary or entitled)
* No understanding of French

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children admitted to hospital pediatric emergencies in France during the pandemic period.
Sampling Method: Non-Probability Sample
Enrollment: 901 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of positivity of COVID-19 virus measured by rt-PCR | At 28 days

SECONDARY OUTCOMES:
Prevalence of positivity of COVID-19 virus measured by rt-PCR in the following subpopulations of emergency patients | at the end an average 28 days
  children admitted to pediatric emergencies for respiratory signs
  * Children hospitalized as a result of travelling to pediatric emergency departments for respiratory signs
  * Respiratory asymptomatic children admitted to pediatric emergencies
Respiratory signs of children tested within 28 day | through study completion, an average 28 days
Percentage of children hospitalized tested within 28 day | through study completion, an average 28 days
Contact frequency | At inclusion
  the degree of relationship with these contacts and the time spent in contact with them within 24 hours before emergency
Prevalence of positivity of other respiratory viruses measured by rt-PCR | at 28 days

CONTACTS AND LOCATIONS:
Overall Officials: François Dubos, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (6):
- France (6):
  - CH Louis MOURIER, Colombes
  - Hôpital Jeanne de Flandres, CHU, Lille
  - Hôpital Mère Enfant CHU, Nantes
  - Hôpitaux Pédiatriques de Nice CHU-Lenval, Nice
  - Hôpital des enfants - CHU, Toulouse
  - CHU de Tours, Tours